CLINICAL TRIAL: NCT02270593
Title: ADAMTS, Proteoglycan and Oxidant / Antioxidant Enzyme Levels of Placenta Previa Totalis(Accreta, Increta, Percreta)
Brief Title: ADAMTS,Proteoglycan and Oxidant / Antioxidant Enzyme Levels of Placenta Previa Totalis (Accreta, Increta, Percreta).
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, sibel özler, ADAMTS, Proteoglycan and Oxidant / Antioxidant Enzyme Levels of Placenta Previa Totalis(Accreta, Increta, Percreta), Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: prospective study-2
Record Dates: First submitted 2014-08-22; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: None Retained — serum and fetal membranes (placenta) and maternal myometrial sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Placenta previa: first; maternal serum, fetal membranes (placenta) and maternal myometrial samples will be investigated for ADAMTS, Proteoglycans and oxidative/antioxidative enzyme status levels in patients with placental invasion anomalies Placenta Previa totalis by ELISA, western blot, immunohystochemistry and PCR (polymerase chain reaction).

SUMMARY:
Placenta previa totalis (accreta, increta, percreta); ADAMTS and proteoglycans and the oxidant / antioxidant enzyme levels.

DETAILED DESCRIPTION:
Placenta previa totalis (accreta, increta, percreta) of pregnant women in the maternal serum, fetal membranes (placenta) and hysterectomy of women with myometrial strips measured the ADAMTS and proteoglycans expression levels, and the oxidant / antioxidant enzyme levels.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women diagnosed with placenta previa by obstetric ultrasound and doppler

Exclusion Criteria:

* Pregnant women with comorbid diseases other than previa totalis .

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: tertiary health institutions
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
ADAMTS,Proteoglycan and Oxidant / Antioxidant Enzyme Levels of maternal serum in patients with the diagnosis of Placenta Previa (Accreta, increta, percreta) | Up to 6 months

SECONDARY OUTCOMES:
ADAMTS,Proteoglycan and Oxidant / Antioxidant Enzyme Levels of myometrial samples in patients with the diagnosis of Placenta Previa (Accreta, increta, percreta) | Up to 6 months
ADAMTS,Proteoglycan and Oxidant / Antioxidant Enzyme Levels of Fetal Membranes in patients with the diagnosis of Placenta Previa (Accreta, increta, percreta) | Up to 6 months
placenta previa totalis in the development, progression and in exacerbating; ADAMTS and proteoglycans, to determine the relationship of changes in expression. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: ahmet nuri danısman, md, Study Director — zekai tahir burak women's health education and research hospital
Locations (1):
- Zekai Tahir Burak Women's Health Education and Research Hospital, Ankara, Turkey (Türkiye)